CLINICAL TRIAL: NCT02827747
Title: The Role of Antioxidants in Keratoconus Patients-A Randomized Controlled Trial of Oral Supplementation of Glutathione, Vitamin A, Vitamin C and Vitamin E
Brief Title: The Role of Antioxidant Supplementation in Keratoconus Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Not enough participant interest.
Sponsor: University of Miami (Other)
Collaborators: Fight for Sight (Other)
Responsible Party: Principal Investigator, Ellen Koo, Assistant Professor of Ophthalmology, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20150646
Record Dates: First submitted 2016-02-25; First posted 2016-07-11 (Estimated); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Keratoconus
Keywords: Keratoconus progression; Vitamins and keratoconus; Vitamin supplementation
MeSH Terms: conditions — Keratoconus | interventions — Antioxidants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo with Dietary Sources of Vitamins (Placebo Comparator): Persons assigned to placebo, who obtain Vitamins A, C, E and Glutathione from dietary sources alone, and have not been on oral RDA supplementation, in the 1 month leading up the time of enrollment and throughout the study period.
  Interventions: Other: Placebo; Combination Product: Dietary Sources
- Antioxidants(Vitamins A,C,E) plus GSH, plus Centrum (Active Comparator): Persons assigned to the study medication, and are continuing the take an oral RDA supplementation, in the form of Centrum.
  Interventions: Other: Antioxidants (Vitamins A,C,E) plus GSH; Dietary Supplement: Centrum
- Antioxidants (Vitamins A,C, E) plus GSH (Active Comparator): Persons assigned to the study medication alone, without oral RDA supplementation in the 1 month leading up the time of enrollment and throughout the study period.
  Interventions: Other: Antioxidants (Vitamins A,C,E) plus GSH
- Placebo plus Centrum (Active Comparator): Persons assigned to placebo, who have been on oral RDA supplementation, who would continue to do so throughout the study.
  Interventions: Other: Placebo; Dietary Supplement: Centrum

INTERVENTIONS:
Other: Antioxidants (Vitamins A,C,E) plus GSH — Study medication would contain 500 milligrams of vitamin C, 400 International Units of vitamin E, and 15 milligrams of beta-carotene (the equivalent to 25,000 International Units of vitamin A).The study medication would also contain 1000mg of Glutathione (GSH).
  Arms: Antioxidants (Vitamins A,C, E) plus GSH; Antioxidants(Vitamins A,C,E) plus GSH, plus Centrum
Other: Placebo — Placebo pill
  Arms: Placebo plus Centrum; Placebo with Dietary Sources of Vitamins
Dietary Supplement: Centrum — Centrum
  Arms: Antioxidants(Vitamins A,C,E) plus GSH, plus Centrum; Placebo plus Centrum
Combination Product: Dietary Sources — From dietary sources of vitamins.
  Arms: Placebo with Dietary Sources of Vitamins

SUMMARY:
Keratoconus is the most common primary cornea ectasia, where the cornea undergoes structural changes, leading to loss of tissue integrity and vision loss. The prevalence of Keratoconus is 1:2000 in the general population. Oxidative stress has been thought to have a major effect in the disease pathogenesis of Keratoconus. In vitro studies have shown increase in metabolites related to oxidative stress in Keratoconus disease, and that Keratoconus cells undergo increased oxidative stress and tissue damage. Animal models have shown a therapeutic effect of Vitamin C (ascorbate) in corneal wound healing. Glutathione and Vitamins A, C, and E are important antioxidants in the human body. To this date, the role of systemic antioxidant supplementation in Keratoconus patients has yet to be studied. In addition, it has yet to be established as to whether there is a correlation between serum antioxidant levels, and the severity of disease in the Keratoconus patient. The investigators propose to investigate the plasma levels of antioxidants in relation to disease severity. The investigators will also investigate the role of antioxidant supplementation-consisting of parenteral Glutathione (GSH), and Vitamins A, C and E-in delaying the disease progression in Keratoconus.

ELIGIBILITY:
Inclusion Criteria:

* Participants would be without illness or condition that could make follow-up, or compliance with study medication difficult.
* Participants may have a prior diagnosis of Keratoconus, or may be diagnosed at the initial visit.
* Participants should not have an eye diagnosis, other than Keratoconus, that could adversely influence the visual acuity.
* These participants must not have had prior surgical procedure to treat Keratoconus, including collagen cross-linking, Intacs ring segments, or corneal transplantation.

Exclusion Criteria:

* would exclude smokers and former-smokers.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Acuity Measured by Snellen Chart | Baseline to 24 months

SECONDARY OUTCOMES:
Change in cornea thickness as measured by video keratography | Baseline to 24 months
Plasma level of Vitamin A | Baseline to 24 months
  Blood draws to look at plasma level of Vitamin A
Plasma level of Vitamin C | Baseline to 24 months
  Blood draws to look at plasma level of Vitamin C
Plasma level of Vitamin E | Baseline to 24 months
  Blood draws to look at plasma level of Vitamin E
Plasma level of Glutathione (GSH) | Baseline to 24 months
  Blood draws to look at plasma level of GSH

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Koo, M.D., Principal Investigator — University of Miami
Locations (1):
- Bascom Palmer Eye Institute-- Palm Beach Gardens, Palm Beach Gardens, Florida, United States

IPD SHARING:
Plan to Share IPD: No